CLINICAL TRIAL: NCT03120793
Title: Assessing Pleural Pressure Changes Between Supine, Upright and Prone Mechanical Ventilation
Brief Title: ARDS Esophageal Balloon Pressure Changes With Positioning Study
Status: Terminated | Type: Observational
Why Stopped: Failure to recruit/enroll
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0135
Record Dates: First submitted 2017-03-20; First posted 2017-04-19 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: ARDS; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Esophageal balloon catheter placement: This is the primary and only arm of the study in which acute respiratory distress syndrome patients will have an esophageal balloon catheter placed with pressures recorded in the supine, upright and prone positions
  Interventions: Device: Esophageal balloon catheter

INTERVENTIONS:
Device: Esophageal balloon catheter — Measurements obtained from mechanically ventilated patients with ARDS in the supine, upright and prone positions

SUMMARY:
The use of esophageal balloon catheters, which use esophageal pressure as a surrogate measurement for transpleural pressure, shows promise in improving outcomes of patients with severe acute respiratory distress syndrome (ARDS) requiring mechanical ventilator. The investigators hope to measure changes in in transpleural pressures in patients undergoing treatment with mechanical ventilation while switching from the supine, upright (head of bed >30 degrees), and prone positions. The goal will be to measure the changes in chest wall and lung compliance in mechanically ventilated patients with changes in position.

DETAILED DESCRIPTION:
The use of esophageal balloon catheters shows promise in improving outcomes of patients with severe ARDS. The estimation of pleural pressure (Ppl) has been validated in the upright position in humans with few studies commenting on the changes in supine positioning and almost none on prone positioning aside from radiographic analysis. An abstract presented at the annual American Thoracic Society meeting recently reported a series of 18 patients undergoing spinal surgery. In this population of patients without ARDS, esophageal pressure (Pes) decreased when shifting from supine to prone positioning. This suggests that transpleural pressure (PtmL) would be increased at a given airway pressure.

The investigators hope to measure changes in PtmL in patients undergoing treatment with mechanical ventilation while switching from the supine, upright (head of bed >30 degrees), and prone positions. The esophageal balloon catheter will be placed using standard techniques and secured with tape to the patients' nares during changes in positioning. The goal will be to measure the changes in chest wall and lung compliance in mechanically ventilated patients with changes in position.

ELIGIBILITY:
Inclusion Criteria:

* age at least 18 years old, need for mechanical ventilation, moderate or severe ARDS, and the ability to tolerate prone positioning.

Exclusion Criteria will be patients who:

* are deemed too ill by their clinicians to be included in the study
* have esophageal or nasopharyngeal pathology (such as tumors, sinusitis, epistaxis, ulcerations, recent surgery or bleeding varices) preventing insertion of the esophageal balloon catheter
* diverticulitis
* bronchopulmonary fistula
* solid-organ transplantation
* history of difficult intubation or airway management
* or contraindications to prone positioning (per the UNC Medical Intensive Care Unit Pronation Therapy protocol, attached)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients admitted to the medical intensive care unit with moderate to severe ARDS who are candidates for prone ventilation therapy and have no contraindications for the placement of an esophageal balloon catheter.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Esophageal pressure measurements from upright to prone position | Measurements will be obtained in the baseline upright position and repeated after about 4 hours in the prone position.
  Obtained from esophageal balloon catheter measurements in prone and upright positions
Change in Esophageal pressure measurements from upright to supine position | The patient is upright at baseline where measurements will be obtained. About 5 minutes will be spent in the supine position.
  Obtained from esophageal balloon catheter measurements in upright and supine positions

SECONDARY OUTCOMES:
Change in Transmural pressure measurements from upright to prone position | Measurements will be obtained in the baseline upright position and repeated after about 4 hours in the prone position.
  Obtained from combination of esophageal balloon catheter measurements and mechanical ventilator in upright and prone positions
Change in Transmural pressure measurements from upright to supine position | The patient is upright at baseline where measurements will be obtained. About 5 minutes will be spent in the supine position.
  Obtained from esophageal balloon catheter measurements in upright and supine positions
Change in Airway pressure measurements from upright to prone position | Measurements will be obtained in the baseline upright position and repeated after about 4 hours in the prone position.
  Obtained from mechanical ventilator in prone and upright positions
Change in Airway pressure measurements from upright to supine position | The patient is upright at baseline where measurements will be obtained. About 5 minutes will be spent in the supine position.
  Obtained from mechanical ventilator in supine and upright positions

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bice, MD, MS, Principal Investigator — UNC Pulmonology and Critical Care
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No